CLINICAL TRIAL: NCT03682380
Title: An Open-Label, Randomized, Multi-panel, Crossover Study to Evaluate the Relative Oral Bioavailability and Food Effect of Seltorexant (JNJ-42847922) After Single-Dose Administration in Healthy Subjects
Brief Title: A Study of Seltorexant (JNJ-42847922) After Single-Dose Administration in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108503; 42847922MDD1011 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — seltorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1: Seltorexant High Dose (Experimental): In Part 1, participants will receive the following treatments: Treatment A: Two low doses of seltorexant tablets (reference formulation), Treatment B: High dose of seltorexant tablet (Test formulation 1), Treatment C: High dose of seltorexant tablet (Test formulation 2), Treatment D: Two low doses of seltorexant tablets (Test formulation 3), Treatment E: Two low doses of seltorexant tablets (Test formulation 4), Treatment F: Two low doses of seltorexant tablets (Test formulation 5), as one of 6 possible treatment sequences on Day 1 in each treatment Periods (Period 1-6). There will be a washout Period of 7 to 14 days from dosing on Day 1 of each treatment period.
  Interventions: Drug: Seltorexant High Dose
- Part 2: Seltorexant High Dose (Experimental): Participants will receive the following treatments: Treatment G: Two low doses of seltorexant tablets (Reference formulation), Treatment H: High dose or two low doses of seltorexant tablet (Test formulation 1), Treatment I: High dose of seltorexant tablet (Test formulation 2), as one of 6 possible treatment sequences on Day 1 in each treatment Periods (Period 1-3). There will be a washout period of 7 to 14 days from dosing on Day 1 of each treatment period.
  Interventions: Drug: Seltorexant High Dose
- Part 3: Seltorexant Low Dose or High Dose (Experimental): Part 3 will have 3 subparts (Part 3A, Part 3B, and Part 3C). In Part 3A and 3B, participants will receive high dose of seltorexant (selected formulation 6) and two low doses of seltorexant (selected formulation 7) respectively in a different food conditions on Day 1 in each treatment Periods (Periods 1-5). In Part 3C, participants will receive high dose of seltorexant (selected formulation 6) and two low doses of seltorexant (selected formulation 7 ) on Day 1 in each period (Period 1 and 2). There will be a washout period of 7 to 14 days from dosing on Day 1 of each treatment period.
  Interventions: Drug: Seltorexant High Dose; Drug: Seltorexant Low Dose

INTERVENTIONS:
Drug: Seltorexant High Dose — In Part 1, Part 2, and Part 3 (3A and 3C), Seltorexant high dose (either a high dose tablet or two low dose tablets) will be administered orally.
  Other Names: MIN-202; JNJ-42847922
Drug: Seltorexant Low Dose — In Part 3 (3B and 3C), Seltorexant low dose will be administered orally.
  Other Names: MIN-202; JNJ-42847922
  Arms: Part 3: Seltorexant Low Dose or High Dose

SUMMARY:
The purpose of this study is to compare the rate and extent of absorption (relative bioavailability) of seltorexant Phase 3 test formulation(s) relative to a reference Phase 2b tablet formulation dosed in the evening under fasted and semi-fasted conditions (3 hours after meal); to assess the effect of type and timing of the meal on the rate and extent of absorption of seltorexant Phase 3 tablet formulation (low dose and high dose strength) in healthy male and female participants; and to assess the pharmacokinetic of single-dose administration of low dose and high dose of seltorexant in healthy male and female participants 3 hours after meal.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy on the basis of medical history (screening only), physical examination, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and Day 1 (predose)
* Be healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* All female participants (regardless of childbearing potential), must have a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening and a negative urine pregnancy test on Day -1 of each treatment period
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 1 month after the last study drug administration
* A man, who is sexually active with a woman of childbearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the investigator (for example, abstinence, vasectomy, barrier method, partner using effective contraception)

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic (Child-Pugh Score greater than or equal to [>=] 7) or renal insufficiency (estimated glomerular filtration rate [eGFR] less than [<] 60 milliliter per minute per 1.73 meter square [mL/min/1.73m^2] based on the modified diet renal disease [MDRD] formula at screening only), thyroid disease, neurologic (including seizure disorders) or psychiatric disease (depression or anxiety disorder in remission is acceptable), infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results. Significant past gastrointestinal medical history, or any disease/surgery that would with interfere drug absorption
* Clinically significant abnormal values for hematology, clinical chemistry (including thyroid stimulating hormone [TSH] at screening only) or urinalysis at screening or at admission to the study site. It is expected that laboratory values will generally be within the normal range for the laboratory, though minor deviations, which are not considered to be of clinical significance to the investigator, are acceptable
* Clinically significant abnormal physical examination, vital signs, or 12-lead ECG at screening or at admission to the study site though minor deviations, which are not considered to be of clinical significance to the investigator are acceptable
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, oral contraceptives, and hormonal replacement therapy within 14 days before the first dose of the study drug is scheduled. Or has used any systemic herbal medications or dietary supplements including products containing Hypericum perforatum (for example, St. John's Wort) from 21 days before the first dose of study drug is scheduled
* Received a known inhibitor of Cytochrome P450 3A4 (CYP3A4) or CYP2C9 activity within 14 days or a period less than 5 times the drugs half-life; whichever is longer, before the first dose of the study drug is scheduled

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Predose up to 48 hours postdose
  Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve from the Time of Dosing to the Last Measurable Plasma Concentration (AUC[0-last]) | Predose up to 48 hours postdose
  AUC(0-last) is the area under the plasma concentration-time curve from the time of dosing to the last measurable plasma concentration.
Area Under the Plasma Concentration-Time Curve Extrapolated to Infinite Time (AUC[0-infinity]) | Predose, up to 48 hours postdose
  AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated using the observed value of the last non-zero plasma concentration.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Part 1: approximately 16 weeks; Part 2: approximately 10 weeks; Part 3: approximately 39 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Dose-Proportionality of Seltorexant Based on Cmax | Predose up to 48 hours postdose
  Dose proportionality of single doses of low dose and high dose of seltorexant from the Cmax will be assessed.
Dose-Proportionality of Seltorexant Based on AUC(0-last) | Predose up to 48 hours postdose
  Dose proportionality of single doses of low dose and high dose of seltorexant from the AUC(0-last) will be assessed.
Dose-Proportionality of Seltorexant Based on AUC(0-infinity) | Predose up to 48 hours postdose
  Dose proportionality of single doses of low dose and high dose of seltorexant from the AUC(0-infinity) will be assessed.
Plasma Protein Binding (PPB) of Seltorexant and Its Metabolites (M12 and M16) | Predose up to 12 hours postdose
  Plasma protein binding (PPB) of seltorexant and its metabolites (M12 and M16) will be determined by using a qualified liquid chromatography coupled with tandem mass spectrometry (LC-MS/MS) method.
Change from Baseline in Karolinska Sleepiness Scale (KSS) Score | Baseline, Day 1, and Day 2
  The KSS is a self reported, assessment of level of drowsiness at the time of scale administration. This scale is focused mainly on the propensity to fall asleep and has a high validity in measuring sleepiness. It consists of a 9-point Likert scale with response options from: 1=extremely alert, 2=very alert, 3=alert, 4=rather alert, 5=neither alert nor sleepy, 6= some signs of sleepiness, 7=sleepy (but no effort to keep awake), 8= sleepy, some effort to keep awake , 9=very sleepy (fighting sleep).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRAHS, Salt Lake City, Utah, United States